CLINICAL TRIAL: NCT04870619
Title: FOCUSED INTENSIVE REPETITIVE STEP TRAINING - Long-term Follow-up of High Intensity Stepping Training After Stroke in Oslo (FIRST-Oslo - Long-term)
Brief Title: FIRST-Oslo Long-term Follow-up
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Indiana University School of Medicine (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other); City of Oslo (Unknown); Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Bø, Physiotherapist PhD, Oslo University Hospital
Other Study IDs: 216346
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: High Intensity Gait Training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High Intensity Gait Training — The intervention provided in this project is routinely delivered as a standard of care at the participating sites for patients after stroke that have a goal of walking improvement. The intervention consists of 45-60 minute, physical therapy sessions that occur five days per week (not weekends), focusing on prioritizing stepping practice at higher aerobic intensities during scheduled treatments (target training zone of 70-85% heart rate max (HRmax). Stepping is performed on treadmills and over ground, with safety harness systems and body weight support only as needed to ensure successful stepping. Tasks are progressed by increasing task difficulty as determined by the therapist. Accordingly, practice of non-walking tasks performed during physiotherapy, including bed mobility, transfers, and standing balance/ pre-gait activities, is limited.

SUMMARY:
The study aims to describe the functional level of the patients who received high intensity gait training during inpatient stroke rehabilitation at discharge, three, six and twelve months after stroke. These data will determine if the observed gains from the high-intensity gait training are retained after discharge from inpatient rehabilitation.

DETAILED DESCRIPTION:
The study is a cohort-study that will have a prospective observational design. This design allows us to follow patients who presently have had a stroke and received high intensity stepping training over time. At this time little is known about the patient's functional trajectory the first 12 months after receiving high intensity stepping treatment as no study has examined long-term effects of high-intensity stepping training delivered in inpatient rehabilitation for stroke in Norway nor internationally.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old) who are receiving inpatient rehabilitation for stroke
* < six months post-stroke
* have the goal to improve walking function
* provide written consent will participate in the study.

Exclusion Criteria:

* inability to consent
* use of bracing or instrumentation (e.g. ventilator) that limits walking
* independence in walking outdoors and on stairs (Functional Ambulation Category (FAC) at admission = 5)
* uncontrolled cardiopulmonary, metabolic, infectious or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two separate inpatient rehabilitation units in Oslo will participate in the study - OUH's rehabilitation unit and OMS' rehabilitation unit, both at Aker campus.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
10 meter walk test | 12 months
  Walking speed
6-minute walk test | 12 months
  Walking distance
Berg balance scale | 12 months
  Balance measured on a scale 0-56 points, higher scores mean a better outcome
Steps | Daily through stay, average of 3 weeks
  Number of Steps
Intensity | Each PT session trough stay, and average of 3 weeks
  Heart Rate during training

SECONDARY OUTCOMES:
Sit-to-stand x5 | 3 weeks
  Functional strength, time to complete in sec
Sit-to-stand x5 | 3 months
  Functional strength, time to complete in sec
Sit-to-stand x5 | 6 months
  Functional strength, time to complete in sec
Sit-to-stand x5 | 12 months
  Functional strength, time to complete in sec
Manual muscle testing | 3 weeks
  Strength of lower extremities, ordinal scale 0-5, higher score indicate better outcome
Manual muscle testing | 3 months
  Strength of lower extremities, ordinal scale 0-5, higher score indicate better outcome
Manual muscle testing | 6 months
  Strength of lower extremities, ordinal scale 0-5, higher score indicate better outcome
Manual muscle testing | 12 months
  Strength of lower extremities, ordinal scale 0-5, higher score indicate better outcome
Action-Research-Arm-Test (ARAT) | Weekly during inpatient stay, in average 3 weeks
  Evaluation tool for motot function in the upper extremity after neurological injuries. Ordinal scale 0-57, higher score indicate better outcome
Action-Research-Arm-Test (ARAT) | 3 weeks
  Evaluation tool for motot function in the upper extremity after neurological injuries. Ordinal scale 0-57, higher score indicate better outcome
Action-Research-Arm-Test (ARAT) | 3 months
  Evaluation tool for motot function in the upper extremity after neurological injuries. Ordinal scale 0-57, higher score indicate better outcome
Action-Research-Arm-Test (ARAT) | 6 months
  Evaluation tool for motot function in the upper extremity after neurological injuries. Ordinal scale 0-57, higher score indicate better outcome
Action-Research-Arm-Test (ARAT) | 12 months
  Evaluation tool for motot function in the upper extremity after neurological injuries. Ordinal scale 0-57, higher score indicate better outcome
EQ-5D-5L | 3 weeks
  Health related quality of life
EQ-5D-5L | 3 months
  Health related quality of life
EQ-5D-5L | 6 months
  Health related quality of life
EQ-5D-5L | 12 months
  Health related quality of life
PROMIS | 3 weeks
  Health related quality of life
PROMIS | 3 months
  Health related quality of life
PROMIS | 6 months
  Health related quality of life
PROMIS | 12 months
  Health related quality of life
10 meter walk test | Weekly through stay, average of 3 weeks
  Walking speed, time in m/sec
10 meter walk test | 3 weeks
  Walking speed, time in m/sec
10 meter walk test | 3 months
  Walking speed, time in m/sec
10 meter walk test | 6 months
  Walking speed, time in m/sec
6 minute walk test | Weekly through stay, average of 3 weeks
  Walking distance in meters
6 minute walk test | 3 weeks
  Walking distance in meters
6 minute walk test | 3 months
  Walking distance in meters
6 minute walk test | 6 months
  Walking distance in meters
Berg balance scale | Weekly through stay, average of 3 weeks
  Balance measured on a scale 0-56 points, higher scores indicate a better outcome
Berg balance scale | 3 weeks
  Balance measured on a scale 0-56 points, higher scores indicate a better outcome
Berg balance scale | 3 months
  Balance measured on a scale 0-56 points, higher scores indicate a better outcome
Berg balance scale | 6 months
  Balance measured on a scale 0-56 points, higher scores indicate a better outcome
MiniBESTest | Weekly through stay, average of 3 weeks
  Balance measured on a scale 0-28, higher scores indicate a better outcome
MiniBESTest | 3 weeks
  Balance measured on a scale 0-28, higher scores indicate a better outcome
MiniBESTest | 3 months
  Balance measured on a scale 0-28, higher scores indicate a better outcome
MiniBESTest | 6 months
  Balance measured on a scale 0-28, higher scores indicate a better outcome
MiniBESTest | 12 months
  Balance measured on a scale 0-28, higher scores indicate a better outcome
Patient Satisfaction with treatment | 12 months
  6 questions on satisfaction with treatment, Likert scale,

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bø, PhD, Principal Investigator — Oslo Univeristy Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Oslo municipality - Enhanced Rehabilitation Aker, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moore JL, Nordvik JE, Erichsen A, Rosseland I, Bo E, Hornby TG; FIRST-Oslo Team. Implementation of High-Intensity Stepping Training During Inpatient Stroke Rehabilitation Improves Functional Outcomes. Stroke. 2020 Feb;51(2):563-570. doi: 10.1161/STROKEAHA.119.027450. Epub 2019 Dec 30. PMID 31884902